CLINICAL TRIAL: NCT02697435
Title: Patient-Centered Versus Imaging-Directed Care for Older Veterans With Chronic LBP
Brief Title: Making Better Lives: Patient-Focused Care for Low Back Pain (LBP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2021-P; PRO 1653 (Other Grant/Funding Number: RR&D)
Record Dates: First submitted 2016-02-12; First posted 2016-03-03 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Chronic Low Back Pain; Hip Ostearthritis; Myofascial Pain Syndrome; Fibromyalgia; Depression; Maladaptive Coping; Lumbar Spinal Stenosis; Insomnia; Sacroiliac Joint Pain; Lateral Hip and Thigh Pain; Anxiety; Dementia; Recent Leg Length Discrepancy
Keywords: Chronic Low Back Pain; Aged; Elderly; Primary Care; Assessment; Lumbar; Spinal Stenosis; Hip Osteoarthritis; Myofascial Pain Syndrome; Fibromyalgia; Depression; Maladaptive Coping; Lumbar Spinal Stenosis; Insomnia; Sacroiliac Joint Pain; Lateral Hip and Thigh Pain; Anxiety; Dementia; Recent Leg Length Discrepancy
MeSH Terms: conditions — Myofascial Pain Syndromes; Fibromyalgia; Depression; Spinal Stenosis; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Dementia; Osteoarthritis, Hip | interventions — Patient-Centered Care

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research Coordinators who perform the "data measure" portion of the baseline are masked from knowing which group (usual care or patient care) the participant ends up in. This is also true of monthly follow-up calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient-Centered Care (Experimental): Patient-centered care will be directed by geriatricians who have been trained to assess and treat 11 conditions that commonly affect chronic low back pain.
  Interventions: Other: Patient-Centered Care
- Imaging-Directed Care (Placebo Comparator): Imaging-Directed Care will allow patients to follow-up their initial imaging with whatever course they (and/or their doctor) chose, should they chose to follow any course at all.
  Interventions: Other: Imaging-Directed Care

INTERVENTIONS:
Other: Patient-Centered Care — Patient-centered care will be directed by geriatricians who have been trained to assess and treat 11 conditions that commonly affect chronic low back pain. Treatments may involve behavioral components, physical therapy, or medical treatments such as cortisone shots, depending on the patient's needs.
  Arms: Patient-Centered Care
Other: Imaging-Directed Care — Imaging-Directed Care will allow patients to follow-up their initial imaging with whatever course they (and/or their doctor) chose, should they chose to follow any course at all.
  Arms: Imaging-Directed Care

SUMMARY:
Back pain is a huge problem for millions of Americans, including nearly 11 million Veterans. Our older Veterans suffer the most. Citizens spend billions of dollars, yet consistently get poor results. Primary Care Providers are often tasked with diagnosing and treating Chronic Low Back Pain, even though they are often undereducated in the field. These PCPs often use advanced imaging, usually MRIs to guide care. These images often show degenerative disc disease and other common pathologies in older adults, even those who are pain free, which can lead to misdiagnosis and treatment. The investigators believe that Chronic Low Back Pain is a syndrome, a final common pathway for the expression of multiple contributors that often lie outside the spine itself. For example, hip osteoarthritis, knee pain, and even anxiety could all lessen back pain if addressed and treated probably.

Investigators will measure participants' low back pain-associated disability with the well-validated RMDQ. Data will be collected at baseline and monthly via telephone. The investigators hypothesize that veterans who receive PCCET will experience significantly greater reduction in low back pain-associated disability than those who receive IAUC at six months.

Investigators will also measure participants' low back pain with the 0-10 Numeric Rating Scale for Pain. Data will be collected at baseline and monthly via telephone. The investigators hypothesize that veterans who receive PCCET will experience significantly greater reduction in low back pain than those who receive IAUC at six months.

The goal of this study is to compare patients treated with usual care, which usually starts with imaging, versus patients who are treated by trained geriatricians who know how to recognize and address 11 key conditions that commonly drive pain and disability in older adults. The investigators believe that older patients who receive care tailored to their needs by educated PCPs will ultimately have less back pain and, more importantly, better quality of life.

DETAILED DESCRIPTION:
Nearly half of our 22 million US military Veterans are age 65 and older and, within this population, low back pain is common, costly and often disabling. The prevalence of low back pain in those 85+, the most vulnerable and fastest growing segment of society, is estimated at 44%. Chronic low back pain (CLBP, i.e., present for 6 months or more) is associated with the overwhelming majority of healthcare resource utilization and personal suffering. Treating back problems cost Americans more than $30 billion in 2007- up from $16 billion in 1997 (in 2007 dollars). Despite these staggering data, there is no evidence that the care of patients with CLBP has improved, and the use of invasive, potentially morbid, and often ineffective interventions (e.g., epidural corticosteroid injections and spine surgery) continues to skyrocket. Primary care providers (PCP) who are tasked with treating CLBP without adequate education often use advanced imaging (most commonly magnetic resonance imaging [MRI]) to guide care. Imaging-identified pathology (e.g., degenerative disc and facet disease, bulging discs) is ubiquitous in older adults, even in those that are pain-free. It is not surprising, therefore, that imaging-guided treatments often lead to suboptimal outcomes and potential morbidity. In contrast to how CLBP is often conceptualized and treated, the investigators conceptualize CLBP as a syndrome, that is, a final common pathway for the expression of multiple contributors that often lie outside the spine itself, for example, hip osteoarthritis, fibromyalgia syndrome, and anxiety. Treating CLBP and ameliorating disability in older adults necessitates addressing multiple conditions and risk factors; however, the expertise to evaluate and treat all of the disorders that can contribute to CLBP typically resides in multiple specialty silos, making a comprehensive approach to treating CLBP difficult to implement.

Through the support of a 2-year Rehab R&D Merit Review pilot award, the investigators have laid the essential foundation for delivering more comprehensive and patient-centric care to older Veterans with CLBP. The investigators have:

* 1) synthesized, through a modified Delphi process, evidence on evaluating and treating 11 key conditions that commonly drive pain and disability in older adults with CLBP
* 2) created algorithms to be used in the clinical setting to treat these 11 conditions
* 3) successfully trained geriatrician providers in a practical structured assessment of the 11 conditions, and
* 4) validated the prevalence of these conditions specifically in older Veterans

In the current application, the investigators are proposing a 2-site pilot study to explore the impact of delivering patient-centered comprehensive evaluation and treatment (PCCET) as compared with imaging-associated usual care (IAUC) to older Veterans with CLBP. In addition to examining whether PCCET is more effective than IAUC for reducing pain and functional limitations when delivered by geriatricians in 2 VA medical centers, the investigators will evaluate PCCET's impact on health-related quality of life and health care utilization. The investigators also will collect data to identify barriers and facilitators to implementing PCCET from the perspective of patients and providers.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking (to ensure the validity of data collected)
* Age 60 and older
* Lumbar MRI within past 30 days and is without evidence of infection, malignancy, or acute fracture OR scheduled for a lumbar MRI within the next 30 days
* CLBP, defined as pain in the lower back of at least moderate severity (assessed with a verbal rating scale), every day or almost every day, for at least 3 months
* No red flags that would indicate a serious underlying disorder that would necessitate urgent and specialized treatment, i.e.,

  * weight loss
  * fever
  * sudden severe LBP
  * change in bowels/bladder
  * back pain that awakens from sleep
  * recent leg weakness
* No pain in other body locations that is more severe than their low back pain
* No psychotic symptoms
* No previous spine surgery
* No dementia (Folstein Mini-Mental State Examination score of > 24)
* No acute illness
* No prohibitive communication impairment (e.g., severe hearing or visual impairment)
* Able to commit to 6 months of study participation

Exclusion Criteria:

* Vulnerable subjects will not be enrolled
* Neither pregnant subjects nor women of childbearing potential will be included because the investigators are targeting older Veterans with CLBP
* Neither children nor prisoners will be included
* Incompetent subjects will be excluded from participating in this research, as determined by performance on the Folstein Mini Mental State Examination

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Weiner, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Using an IRB-approved waiver of consent, research coordinators (RCs) screened CPRS records of Veterans age 60-89 with low back pain.Those eligible were mailed a study brochure and a letter signed by the chief of Primary Care. Additional screening was performed on those who called the RC. Those eligible were further screened on site.
Pre-assignment Details: There was no wash out or run in period.
Period: Overall Study
Arm/Group | Patient-Centered Care | Imaging-Directed Care
Started | 25 | 30
Completed | 24 | 26
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-Centered Care | Imaging-Directed Care | Total
Number analyzed (Participants) | 25 | 30 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 12 | 16
  >=65 years | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (7.5) | 67.2 (5.5) | 69.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 24 | 29 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants' Level of Low Back Pain-associated Disability as Assessed by Roland Morris Disability Questionnaire (RMDQ)
Description: The Roland Morris Questionnaire is a 24 item yes/no measure of back pain interference with various daily activities. It is a well validated measure of low back pain disability. The total score ranges from 0 to 24 with a higher score meaning greater impairment. Our main outcome measure is reported as the change in Roland Morris score from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: All participants were called monthly for 6 months. One main outcome measure was Roland Morris score at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patient-Centered Care: Patient-Centered Care (i.e., ABC care): Patient-centered care will be directed by geriatricians who have been trained to assess and treat 11 conditions that commonly affect chronic low back pain in older adults. Treatments may involve behavioral components, physical therapy, or medical treatments such as cortisone shots, depending on the patient's needs.
Arm/Group | Patient-Centered Care | Imaging-Directed Care
Number analyzed (Participants) | 24 | 26
score on a scale | -1.29 (6.05) | -0.08 (4.12)
Statistical Analysis 1: Comparison: Patient-Centered Care vs Imaging-Directed Care; Test type: Superiority; p < 0.05, Mixed Models Analysis — P-value is calculated

2. Primary Outcome: Participants' Average 7-day Self-reported Level of Low Back Pain as Assessed by 0-10 Numeric Rating Scale
Description: Pain rated on a scale of 0 to 10, where 0 is no pain and 10 is worst possible pain. Outcome is change score.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient-Centered Care | Imaging-Directed Care
Number analyzed (Participants) | 24 | 26
units on a scale | 0.46 (2.99) | 0.96 (2.18)

ADVERSE EVENTS:
Time Frame: through the duration of the study, up to 2 years.
Arm/Group | Patient-Centered Care | Imaging-Directed Care
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/30
Other Adverse Events (participants affected / at risk) | 0/25 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT02697435/Prot_SAP_000.pdf